CLINICAL TRIAL: NCT01126281
Title: THE USE OF FLOSEAL GELATIN MATRIX FOR THE HAEMOSTASIS DURING LAPAROSCOPIC CHOLECYSTECTOMY FOR ACUTE CHOLECYSTITIS; EFFICACY AND SAFETY EVALUATED IN A MULTICENTER, PROSPECTIVE, OPEN LABEL TRIAL WITH AN HISTORICAL CONTROL GROUP. (G.L.A. STUDY: GELATIN Matrix in Laparoscopic Cholecystectomy for Acute Cholecystitis)
Brief Title: Efficacy and Safety of Floseal for the Haemostasis During Laparoscopic Cholecystectomy in Acute Cholecystitis (GLA)
Acronym: GLA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bologna (Other)
Responsible Party: General, Emergency and Transplant Surgery dept., Sant'Orsola Malpighi University Hospital, Bologna, Italy
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sant'orsola1
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2010-05

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cholecystectomy, Laparoscopic

ARMS (1):
- Floseal use (Experimental)
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Laparoscopic cholecystectomy

SUMMARY:
The aim of this study is to evaluate the effect and safety of Floseal in this preliminary prospective trial with patients undergoing acute laparoscopic cholecystectomy for acute cholecystitis

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 - 65
* Clinical (pain, fever > 37.5 °C, WBC > 10.000 / microL), and ultrasound evidence of cholecystitis
* Surgical indication for laparoscopic cholecystectomy
* ASA class I-III
* Informed consent
* <72 hours from onset of symptoms

Exclusion Criteria:

* Informed consent refusal
* Choledocholithiasis
* Pre surgical generalized peritonitis (clinical evaluation)
* ASA class > III
* Peripheral artery disease
* Active or past history of malignant systemic disease
* Pregnant or lactating females
* Known allergy to components Floseal including bovine allergy (bovine gelatin)
* Known drug or alcohol abuse
* Patients with known diabetes, chronic renal disease and other metabolic diseases
* Patients in chronic cortisone treatment more than 2 years before surgery
* Patients on chronic use of platelet inhibitors such as Aspirin, Plavix, NSAID's etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-08; Primary Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
to evaluate the percentage of patients with complete haemostasis 10 minutes after laparoscopic application of haemostatic agent (Floseal) to the gall bladder bed. | 10 minutes

SECONDARY OUTCOMES:
• Percentage of patients with complete haemostasis evaluated at 2, 4 and 6 minutes after laparoscopic application of haemostatic agent (Floseal) to the gall bladder bed. | 6 minutes
• Surgery time. | 3 year
• Percentage of patients with conversion from laparoscopic procedure to open laparotomy (conversion rate). | 3 year
• Percentage of patients developing post operative bleeding leading to re-operation. | 3 year
• Percentage of patients developing post operative bleeding leading to transfusion of blood | 3 year
• Percentage of patients developing post operative biliary leaking. | 3 year
• Time to drain removal. | 3 year
• Mortality. | 3 year
• Length of stay in hospital. | 3 year
• Safety evaluated as number of patients with adverse events and serious adverse events until end of the study. | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Orsola-Malpighi Univesity Hospital, Bologna, Bologna, Italy